CLINICAL TRIAL: NCT06168097
Title: MicroRNAs Dysregulation as Potential Biomarkers for Effective Diagnosis of Endometriosis
Brief Title: The Use of MicroRNAs Dysregulation as Potential Biomarkers for Effective Diagnosis of Endometriosis
Acronym: ENDMET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Endometriosis-01
Record Dates: First submitted 2023-10-21; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis
Keywords: lining of uterus; Diarrhea or constipation during a menstrual period.; Heavy or irregular periods.; Spotting or bleeding between menstrual periods.
MeSH Terms: conditions — Endometriosis; Diarrhea; Menstruation Disturbances; Metrorrhagia | interventions — Laparoscopy; Laparotomy

STUDY DESIGN:
Intervention Model Description: case control study 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of endometriosis and 100 women undergoing surgery for gynaecological disorders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of endometriosis (Experimental): 1. We Will take Both blood and tissue samples used to study them.
  2. We Will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (Surgical profile) before their planned surgery.
  3. Small tissue samples will be taken from the tissue which is surgically excised as a part of treatment.
  4. It will include tissue from inner lining of uterus (endometrium) in all participants and from excised endometriosis tissue in patients with endometriosis.
  Interventions: Procedure: 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of endometriosis; Procedure: women with intraoperative and / or histopathology findings suggestive of endometriosis
- 100 women undergoing surgery for gynaecological disorders other than endometriosis or adenomyosis (No Intervention): . We Will take Both blood and tissue samples used to study them. 2. We Will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (Surgical profile) before their planned surgery.
  3.Small tissue samples will be taken from the tissue which is surgically excised as a part of treatment.
  4. It will include tissue from inner lining of uterus (endometrium) in all participants and from excised endometriosis tissue in patients with endometriosis.

INTERVENTIONS:
Procedure: 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of endometriosis — 1. We Will take Both blood and tissue samples used to study them.
  2. We Will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (Surgical profile) before their planned surgery.
  3. Small tissue samples will be taken from the tissue which is surgically excised as a part of treatment.
  4. It will include tissue from inner lining of uterus (endometrium) in all participants and from excised endometriosis tissue in patients with endometriosis.
  Arms: 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of endometriosis
Procedure: women with intraoperative and / or histopathology findings suggestive of endometriosis — 1. We Will take Both blood and tissue samples used to study them.
  2. We Will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (Surgical profile) before their planned surgery.
  3. Small tissue samples will be taken from the tissue which is surgically excised as a part of treatment.
  4. It will include tissue from inner lining of uterus (endometrium) in all participants and from excised endometriosis tissue in patients with endometriosis.
  Arms: 100 women undergoing surgery (laparoscopy / laparotomy) with presumed diagnosis of endometriosis

SUMMARY:
OBJECTIVES :

1. To investigate the expression pattern of miRNAs operational in inflammation, angiogenesis, hypoxia, apoptosis and cell proliferation in eutopic and ectopic endometrium of patients with endometriosis and normal endometrium of healthy controls.
2. To understand the function of candidate predictive miRNAs for endometriosis by investigating their downstream targets and associated biological pathways.
3. Evaluation of significant outcome of objective 1 in serum samples to establish them as biomarkers.

Study Design:

Case control study. sample size: 200

DETAILED DESCRIPTION:
METHODOLOGY :

1 Investigator will take Both blood and tissue samples used to study them. 2. Investigator will take approximately 3 ml of blood which will be used from the blood sample collected for routine preoperative tests (Surgical profile) before their planned surgery.

3.Small tissue samples will be taken from the tissue which is surgically excised as a part of treatment.

4. It will include tissue from inner lining of uterus (endometrium) in all participants and from excised endometriosis tissue in patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients having more severe forms of endometriosis (Stage III and IV)
* The probands were chosen randomly from the pool of available endometriosis patients and healthy controls of Indian origin.

Exclusion Criteria:

* Diagnosis of non-endometriotic ovarian cysts, adenomyosis, ovarian cancer, fibroids, and stage I and II endometriosis.
* Exclusion criteria defined for the control group were personal history of chronic pelvic pain, secondary dysmenorrhea, abnormal uterine bleeding and family history of endometriosis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
2. To understand the function of candidate predictive miRNAs for endometriosis by investigating their downstream targets and associated biological pathways | 3 years
  ROC curve analysis is to estimate the sensitivity and specificity of miRNA expression levels to establish them as biomarkers for endometriosis.

SECONDARY OUTCOMES:
To investigate the expression pattern of miRNAs and their downstream targets in endometrial tissues (samples of normal adult endometrium and ectopic and eutopic endometrium of patients with endometriosis) | 3 years
  Western Blot and immunohistochemical analysis (IHC) for expression analysis..

CONTACTS AND LOCATIONS:
Overall Officials: Shraddha Ramchandani, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Shraddha Ramchandani, Hyderabad, Telanagana, India

IPD SHARING:
Plan to Share IPD: No